CLINICAL TRIAL: NCT07314502
Title: Prenatal Exercise Including Perineal Massage and Maternal-Neonatal Outcomes: A Randomized Controlled Trial
Brief Title: Prenatal Exercise Including Perineal Massage and Maternal-Neonatal Outcomes
Acronym: PEPM-RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: South China Normal University (Other)
Collaborators: Guangdong Provincial Maternal and Child Health Hospital (Other); Technical University of Madrid (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Dingfeng Zhang, Principal Investigator, South China Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20250094; 20250094 (Other: Guangdong Provincial Maternal and Child Health Hospital)
Record Dates: First submitted 2025-11-21; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Urinary Incontinence; Postpartum Depression (PPD); Neonatal Complications; Gestational Diabetes
Keywords: Exercise; Urinary Incontinence; Postpartum Depression; Macrosomia; Pregnancy
MeSH Terms: conditions — Depression, Postpartum; Diabetes, Gestational; Motor Activity; Urinary Incontinence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants will receive routine prenatal care and a supervised prenatal exercise throughout pregnancy including perineal massage at late pregnancy.
  Interventions: Other: Supervised prenatal exercise including antenatal perineal massage
- Control (No Intervention): Participants will receive routine prenatal care and will not receive the structured supervised exercise program or professionally administered antenatal perineal massage

INTERVENTIONS:
Other: Supervised prenatal exercise including antenatal perineal massage — Following random allocation, pregnant participants will participate in supervised prenatal exercise sessions three times weekly, with each session lasting 60 minutes. From 36 weeks' gestation onward, antenatal perineal massage will be administered by trained healthcare professionals at the hospital.
  Arms: Exercise group

SUMMARY:
The study is divided into three phases:

Phase 1: Baseline survey to obtain an overall understanding of the current situation of voluntary participation in prenatal perineal massage.

Phase 2: Follow-up survey to further assess the current situation of voluntary prenatal exercise and prenatal perineal massage.

Phase 3: Implementation of an intervention combining prenatal exercise and perineal massage.

The goal of this clinical trial is to learn whether a combined prenatal program of supervised, moderate-intensity exercise plus professionally administered antenatal perineal massage can improve maternal and newborn outcomes and can be safely implemented as part of routine antenatal care in healthy pregnant women receiving care at participating hospitals.

The main questions it aims to answer are:

1. Does the combined prenatal program reduce urinary incontinence during pregnancy and after delivery?
2. Does the combined prenatal program reduce depressive symptoms during pregnancy and in the postpartum period?
3. Does the combined prenatal program lower the risk of gestational diabetes mellitus?
4. Does the combined prenatal program reduce neonatal complications, including macrosomia?
5. Do spontaneous, self-initiated prenatal exercise and structured, supervised prenatal exercise differ in their effects on maternal and neonatal outcomes ()?

Researchers will compare the combined prenatal program to usual antenatal care to determine whether the intervention improves maternal and neonatal outcomes and is safe, feasible, and acceptable in a real-world clinical setting.

Participants will:

1. Be screened and enrolled during pregnancy and complete baseline and follow-up assessments during pregnancy and after delivery.
2. Be randomly assigned to either an intervention group or a usual-care control group.
3. If assigned to the intervention group, attend supervised moderate-intensity exercise sessions three times per week (approximately 60 minutes per session) throughout pregnancy and receive antenatal perineal massage delivered by trained health professionals during late pregnancy.
4. Provide questionnaire-based information and clinical data collected during routine visits and from medical records for outcome evaluation.

DETAILED DESCRIPTION:
This project is conducted in a provincial Maternal and Child Health Hospital network (one leading center plus three collaborating hospitals) and is organized into three phases: (1) a baseline survey, (2) a prospective observational follow-up, and (3) a parallel-group randomized controlled trial (RCT) implemented in routine care.

Overall design and procedures Phase 1 uses a cross-sectional baseline survey (planned n=3,000; Nov 25-Dec 31, 2025) to describe current voluntary participation in prenatal perineal massage. Phase 2 is a prospective follow-up cohort (planned n=2,000; Jan 1, 2026-Jan 31, 2028) tracking participants from the first antenatal visit through 24 months postpartum to evaluate real-world patterns of spontaneous prenatal exercise and voluntary perineal massage and their associations with maternal and neonatal outcomes. Phase 3 is a two-arm, parallel-group RCT (planned n=2,000; Jan 1, 2026-Dec 31, 2028) comparing a structured combined prenatal program versus usual antenatal care, with follow-up extended to 36 months postpartum.

Participants and setting Pregnant women receiving routine antenatal care at participating hospitals will be screened by clinical staff. Eligibility and exclusion criteria are provided in the record's Eligibility section. Written informed consent will be obtained prior to any study-specific procedures.

Randomization and masking (Phase 3) In the RCT, participants will be randomized in a 1:1 ratio using a computer-generated allocation sequence managed centrally by designated staff at the leading center. Allocation concealment procedures will be applied for staff involved in outcome assessment and data management when feasible. Due to the nature of the intervention, participants and intervention staff cannot be blinded; however, outcome assessment and data analysis will be performed with masking whenever operationally feasible.

Intervention (Phase 3) Participants assigned to the intervention group will receive (1) a supervised, moderate-intensity prenatal exercise program and (2) professionally administered antenatal perineal massage during late pregnancy.

Exercise program: Sessions will be delivered three times per week, approximately 60 minutes per session, from enrollment through pregnancy. The exercise intervention was conducted at the collaborating hospitals. The exercise program consisted of seven components: warm-up, aerobic exercises, strength training, balance and coordination exercises, stretching and relaxation, pelvic floor muscle training coordinated with breathing (10 sets of slow contractions held for 8-12 seconds each and 3 sets of rapid contractions lasting 25-30 seconds each), and a post-session communication/wrap-up debrief. Exercise intensity will be maintained at a moderate level and adjusted based on gestational age, maternal symptoms, perceived exertion, and available physiological monitoring, following established safety principles for physical activity during pregnancy. Sessions will be delivered individually or in small groups at the hospital or a designated facility.

Perineal massage: During late pregnancy, participants will receive antenatal perineal massage provided by trained health professionals using standardized operating procedures to support consistency and safety.

Comparator (Phase 3) The control group will receive routine prenatal care as provided by participating hospitals, including general health education and standard advice delivered in usual practice. They will not receive the structured supervised exercise sessions or professionally administered perineal massage that define the intervention. Any additional clinical management deemed necessary by treating clinicians will be permitted and recorded.

Intervention delivery, training, and fidelity Intervention delivery staff will receive study-specific training before participant enrollment. Exercise sessions will be supervised by personnel with relevant physical education training backgrounds working under the oversight of clinicians and senior researchers. Standardized materials and monitoring logs (e.g., Attendance will be recorded using a computer-based application) will be used to support implementation fidelity and to document adherence.

Follow-up and data sources Data will be collected at prespecified time points during pregnancy, at delivery, and during postpartum follow-up. Maternal and neonatal outcomes are specified in the Outcome Measures section of the record and will be assessed using validated instruments and clinical information, with delivery and neonatal outcomes extracted from hospital records by trained staff.

Safety monitoring Exercise intensity will be supervised and adjusted to maintain a moderate workload, targeting 55-65% of the maternal maximum heart rate calculated using the Karvonen formula, and corroborated by a Borg Rating of Perceived Exertion score of 12-14 ("Somewhat Hard"). Heart rate will be monitored using a heart rate monitor or wearable activity tracker, with accelerometer-based monitoring used when available to support intensity supervision; when electronic monitoring is not feasible, heart rate will be assessed manually via palpation at the carotid artery. Accelerometers will also be used to monitor the health status of pregnant women.

Data management and analysis overview Data will be recorded using standardized case report forms and entered into a secure database with quality-control procedures (REDCap). The primary analytical approach for the RCT will compare outcomes between groups according to the intention-to-treat principle, consistent with a prespecified statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years；
* Gestational age between 8 and 16 weeks
* No contraindications to exercise；
* Able to attend in-person exercise classes；
* Having obtained hospital approval to participate in this exercise program；
* Able to carry out basic communication in Mandarin Chinese;
* Planning to deliver at the same maternal and child health hospital.

Exclusion Criteria:

* Unable to deliver at the same hospital due to personal reasons；
* Currently participating in other research projects；
* Presence of absolute contraindications to exercise；
* Uncertain about being able to attend three in-person exercise sessions per week；
* Unable to communicate in Mandarin Chinese.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) or Patient Health Questionnaire-9 (PHQ-9) total score | Baseline (after randomization); 28 and 36 weeks' gestation; and 1, 2, 4, 6, 8, 12, 24, 36 months postpartum
  Depressive symptoms score： Depressive symptoms will be assessed using the 1. Edinburgh Postnatal Depression Scale (The scale consists of a total of 10 items, each scored on a four-point Likert scale ranging from 0 to 3, with a maximum total score of 30. A total score greater than 12 is considered a positive screening result, indicating a high likelihood of perinatal depression in pregnant or postpartum women, and professional medical consultation is recommended. Higher total scores indicate more severe depressive symptoms.) ， or 2. Patient Health Questionnaire-9 (The scale consists of 9 items, each of which is scored based on the frequency of symptoms experienced over the past two weeks. Each item is rated on a scale from 0 to 3, resulting in a total score ranging from 0 to 27.
  Interpretation of total scores:
  0-4: No depressive symptoms
  5-9: Possible mild depression
  10-14: Possible moderate depression
  15-19: Possible moderately severe depression
  20-27: Possible severe depress).
Number of participants with urinary incontinence assessed by the International Consultation on Incontinence Questionnaire (ICIQ) | 34 weeks' gestation; and 1, 3, 6, 12, 18, 24, and 36 months postpartum
  Urinary incontinence will be assessed using the International Consultation on Incontinence Questionnaire (In this study, urinary incontinence was defined as experiencing urine leakage at least once per week).
Number of participants diagnosed with gestational diabetes mellitus (GDM) | 24-28 weeks' gestation (routine screening), at any time during pregnancy (up to 40 weeks of gestation) if clinically indicated.
  GDM will be determined using a 75-g OGTT according to prespecified diagnostic criteria (e.g., IADPSG/WHO-recommended thresholds as adopted by the participating hospitals). The outcome will be reported as the number (and percentage) of participants meeting the diagnostic criteria during pregnancy, extracted from hospital laboratory and medical records.
Maternal weight (kg) | Pre-pregnancy (self-reported at baseline); early pregnancy (≤13 weeks' gestation); mid-pregnancy (24-28 weeks' gestation); late pregnancy (34-36 weeks' gestation); and 1, 2, 4, 6, 8, 12, 18, 24, and 36 months postpartum
  Maternal weight will be measured in kilograms using standardized clinical assessments and extracted from antenatal and postpartum medical records. Weight will be reported at each prespecified time point and compared between groups.

SECONDARY OUTCOMES:
Mode of delivery (vaginal, operative vaginal, or cesarean) | At delivery (36-40 weeks' gestation)
  Mode of delivery will be classified based on delivery records as vaginal birth (spontaneous), operative vaginal birth (vacuum or forceps), or cesarean delivery. The outcome will be reported as the number (and percentage) of participants in each category and compared between groups.
Episiotomy rate at delivery | At delivery (36-40 weeks' gestation)
  Episiotomy will be recorded from delivery medical records. The outcome will be reported as the number (and percentage) of participants who undergo episiotomy and compared between groups.
Perineal tear severity (first- to fourth-degree) at delivery | At delivery (36-40 weeks' gestation)
  Perineal tears will be classified according to standard obstetric definitions (first-, second-, third-, or fourth-degree) based on delivery records. The outcome will be reported as the number (and percentage) of participants in each tear grade and compared between groups.
Duration of labor from active phase onset to delivery (hours) | At delivery (36-40 weeks' gestation)
  The duration of labor will be defined as the time from the onset of active labor (cervical dilation ≥ 6 cm with regular uterine contractions) to delivery of the neonate. Time will be extracted from standardized labor and delivery records and reported in hours, then compared between groups.
birth weight and early childhood weight | At birth, and 1, 2, 4, 6, 8, 12, 18, 24, and 36 months of age
  birth weight (kilograms) and early childhood weight (kilograms) will be obtained from measurements using a weighing scale.
newborn height and head circumference | At birth, and 1, 2, 4, 6, 8, 12, 18, 24, and 36 months of age
  Height and head circumference (meters) will be measured using a tape measure

CONTACTS AND LOCATIONS:
Locations (1):
- South China Normal University, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Brik M, Sánchez-Polán M, Farràs A, Hernández-Fleury A, Temprado J, Calero I, Higueras T, Silva C, Zhang D, Carreras E, Barakat R. Maternal and cardiovascular factors related to carotid intima-media thickness during pregnancy: A prospective cohort study. — https://doi.org/10.1016/j.ejogrb.2025.113943
- See also: Sánchez-Polán M, Brik M, Silva-Jose C, Zhang D, Díaz-Blanco MÁ, de la Manzanara PH, Arias AM, Alzola I, Barakat R. Physical activity during pregnancy and depression, anxiety and stress: randomized clinical trials. American Journal of Obstetrics & Gynecol — https://doi.org/10.1016/j.ajogmf.2025.101835
- See also: Zhang D, Sánchez-Polán M, Silva-Jose C, Díaz-Blanco Á, Brik M, Arias AM, Hernando P, Barakat R. Prenatal Exercise Decreases Urinary Incontinence in Late Pregnancy and 3 Months Postpartum: A Randomized Controlled Trial. Medicine and science in sports and — https://doi.org/10.1249/mss.0000000000003597
- See also: Related Info — https://bjsm.bmj.com/content/54/23/1395.abstract
- See also: Related Info — https://www.apunts.org/en-guiding-journey-essential-tools-for-articulo-S2666506924000415